CLINICAL TRIAL: NCT04930874
Title: Cerebral Autoregulation and Severe Coronavirus Disease 19 [CA-COVID]: a Single-center Physiological Study
Brief Title: Cerebral Autoregulation and COVID-19
Acronym: CA-COVID
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low rate of enrollment
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, Spyros D. Mentzelopoulos, Professor of Intensive Care Medicine, National and Kapodistrian University of Athens Medical School, University of Athens
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CA-COVID 196/10-6-2021
Record Dates: First submitted 2021-06-15; First posted 2021-06-18 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: COVID-19 Acute Respiratory Distress Syndrome; COVID-19 Pneumonia
Keywords: COVID-19; Cerebrovascular circulation; Spectroscopy, Near-Infrared
MeSH Terms: conditions — COVID-19 | interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ICU patients with COVID-19 (Experimental): NIRS monitoring will be performed for approximately 90 minutes at 2 mean blood pressure levels (MAP, ie 65-70 mmHg and 95-100 mmHg) within 12-48 hours and 60-84 hours after admission to the ICU for severe COVID-19 infection. Autoregulation will be assessed using Tissue Oxygenation Index values and mean arterial pressure values in a regression analysis and will be considered sufficient if the relative Pearson correlation coefficient is less than 0.3. Cerebral blood flow will be assessed by blood flow index determination after intravenous infusion of 5 mg indocyanine.
  Interventions: Other: NIRS (Near-Infrared Spectroscopy)

INTERVENTIONS:
Other: NIRS (Near-Infrared Spectroscopy) — NIRS assessment of cerebral autoregulation and cerebral blood flow

SUMMARY:
This study aims to assess cerebral autoregulation by near-infrared spectroscopy (NIRS) in patients with severe coronavirus disease 19 (COVID-19). Results on COVID-19 participants will be compared with prior results of patients with septic shock and cardiac arrest, who participated in NCT03649633 and NCT02790788, respectively.

DETAILED DESCRIPTION:
Background and Rationale:

Septic encephalopathy is a serious complication of sepsis / septic shock. In postmortem, human brain samples, two forms of neuraxonal injury have been described, namely, scattered ischemic lesions and diffuse injury. Prior evidence suggests that cerebral autoregulation is impaired in patients with septic shock, and this may render the central nervous system more vulnerable to direct ischemic damage, especially during episodes of hypotension. Recent observational data suggest that impaired cerebral autoregulation is associated with death within 3 months in patients with septic shock. Near-infrared spectroscopy (NIRS) constitutes an established method of noninvasive assessment of cerebral autoregulation and also provides the capability of semiquantitative assessment of regional cerebral blood flow. Severe coronavirus disease (COVID-19) is characterized by hypoxemia due to pneumonia, thromboembolic events that often affect the cerebral and pulmonary vascular network, vasodilatory shock and multiorgan failure. Pathophysiological mechanisms have features in common with those of septic shock and include "cytokine storm", diffuse vascular endothelial involvement, micro- and macro-vascular thrombosis and dysregulation of micro-circulation and vascular tone. In the present study, the following 3 hypotheses will be tested: 1. Cerebral autoregulation is likely to be severely impaired or even abolished in patients with COVID-19 who require admission to an Intensive Care Unit (ICU). In addition, the correlation between the NIRS Tissue Oxygenation Index and the mean arterial pressure may be stronger in COVID-19 compared to septic shock and comparable to that determined after cardiac arrest. 2. Cerebral autoregulation is likely to be associated with known COVID-19 severity markers such as lymphopenia and elevated C-reactive protein (CRP), ferritin, delta dimers (D-dimers) and lactate dehydrogenase (LDH) 3. The early (ie on ICU days 1 and 3) absence of cerebral autoregulation is likely to be associated with residual neurological deficits.

METHODS:

NIRS monitoring will be performed for approximately 90 minutes at 2 mean blood pressure levels (MAP, i.e. 65-70 mmHg and 95-100 mmHg) within 12-48 hours and 60-84 hours after admission to the ICU for severe COVID-19 infection. Autoregulation will be assessed using Tissue Oxygenation Index values and mean arterial pressure (MAP) values in a regression analysis and will be considered sufficient if the relative Pearson correlation coefficient is less than 0.3 Cerebral blood flow will be assessed by blood flow index (BFI) determination after intravenous infusion of 5 mg indocyanine.

ICU Protocol: All COVID-19 patients participating in this study will be treated in a standardized manner that includes: An intermediate dose of Enoxaparin, e.g. 4000 units x 2 subcutaneously 2. Treatment with remdesivir and dexamethasone 3. Up to 2 broad-spectrum antibiotics to treat possibly co-existing bacterial respiratory tract infection 4. A conservative fluid management strategy 5. A protective ventilation strategy in a semirecumbent position 5. Anesthesia with Midazolam, Propofol and Remifentanil 7. Enteral nutrition that will start within 24 hours after admission to the ICU, 8. Permissive hyperglycemia (blood glucose 150-200 mg / dL).

Data Collection and Patient Monitoring:

Monitoring of patients during the first 10 days after inclusion in the study will include 1) Determination and recording of hemodynamic parameters and hemodynamic support, blood gases and arterial blood lactate at 9 p.m. 2) Blood sampling at 24-48, 72 hours and 7 days after inclusion in the study for determination of serum cytokines and 3) Daily recording of laboratory values, fluid balance and administration. The results of 2-4 daily determinations of blood glucose will be recorded and then the incidence of hyperglycemia (defined as blood glucose in excess of 200 mg) will be analyzed. Follow-up until day 60 after inclusion in the study will include organic failures and the number of days without mechanical ventilatory assistance. Finally, the length of stay in the ICU, the date of discharge from the hospital and the morbidity and complications throughout the patient's treatment until discharge from the hospital will be recorded.

Predefined comparisons: The severity of cerebral autoregulation disturbance in patients with COVID-19 will be compared with the cerebral autoregulation disturbance in 1) patients with septic shock (n = 32, NCT03649633, www.clinicaltrials.gov) and 2) cardiac arrest (n = 30, NCT02790788, www.clinicaltrials.gov). Also, other -pre-specified -by the respective research protocols- patient monitoring variables will be compared between the aforementioned groups of patients.

Names / degrees of Associates:

Alexandros Kouvarakos, Physiotherapist; Eirini Patsaki, Physiotherapist; Sotirios Malachias, MD, PhD; Charikleia Vrettou, MD, PhD; Stylianos Kokkoris, MD, PhD; Prodromos Temperikidis, MD, PhD; Aggeliki Kannavou, MD, PhD; George Adamos, MD, PhD

ELIGIBILITY:
Inclusion Criteria:

* Admission to ICU and endotracheal intubation/mechanical ventilation for severe COVID-19 infection

Exclusion Criteria:

* Age <18 years
* Pregnancy
* Patients with a terminal underlying disease who are unlikely to survive until discharge from the hospital
* Patients with acquired immunodeficiency and ("pre-COVID") lymphocyte Cluster Differentiation 4+ count <50 / μL
* Patients with COVID-19 who have been transferred from another hospital
* Patients with a history of allergic reaction
* Use of prone position to facilitate mechanical ventilation
* Absence of signed informed consent from a first degree relative

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2021-06-22 (Actual); Primary Completion 2022-09-16 (Actual); Study Completion 2022-09-16 (Actual)

PRIMARY OUTCOMES:
Cerebral autoregulation | Days 1-4 of ICU admission
  The tissue oxygenation index of the frontal cortex will be determined (at a rate of 180 measurements / min) while increasing MAP from a minimum of 65-75 mmHg to a maximum of 90-100 mmHg by changing the vasopressor infusion rate. Cooncurrent changes in MAP will also be recorded. Subsequently, linear regression between MAP and the Tissue Oxygenation Index will be performed. A Pearson correlation coefficient of >0.3 will be considered as "absence" of autoregulation of the cerebral vasculature.
Cerebral blood flow | Days 1-4 of ICU admission
  Cerebral blood flow at MAP 65-75 mmHg and MAP 90-100 mmHg by determination of the blood flow index.

SECONDARY OUTCOMES:
Neurologic failure free days | Days 1-60 after ICU admission
  Days without neurologic failure throughout the 60-day follow-up period. Patients with a Glasgow Coma Scale of <9 will be considered to have neurological failure.
Ventilator free days | Days 1-60 after ICU admission
  Days without mechanical ventilatory assistance throughout the 60-day follow-up period. On any given day of follow-up, patients will be considered as "ventilator-free" only if there is no need for respiratory support within the preceding 24 hours.
Survival to hospital discharge and neurological outcome | Days 1-60 after ICU admission
  Survival to hospital discharge and neurological outcome assessed by the Cerebral Performance Category Score, and the Modified Rankin Scale Score.
Survival to hospital discharge and neurological outcome | Days 1-60 after ICU admission
  Survival to hospital discharge and neurological outcome assessed by the Cerebral Performance Category (CPC) Score. The CPC Score ranges from 1 to 5, with 1 corresponding to the best possible outcome (i.e. patient able to work and lead a normal life), and 5 corresponding to the worst possible outcome (i.e. brain death).
Survival to hospital discharge and neurological outcome | Days 1-60 after ICU admission
  Survival to hospital discharge and neurological outcome assessed by the Modified Rankin Scale (mRS) Score. The mRS ranges from 0, corresponding to the best possible outcome (i.e. no symptoms related to a neurological deficit), to 6 corresponding to the worst possible outcome (i.e. death).
Serum Cytokines | Days 1-7 after ICU admission
  Tumor Necrosis Factor alpha, Interleukin (IL)-1 beta, IL-6, IL-8, and IL-10 levels at 24-48, 72 hours and 7 days after enrollment. Plasma concentrations of all the aforementioned cytokines will be expressed in picograms per milliliter.

CONTACTS AND LOCATIONS:
Overall Officials: Spyros D Mentzelopoulos, MD, Professor, Principal Investigator — National and Kapodistrian University of Athens; Anastasia D Kotanidou, MD, Professor, Study Chair — National and Kapodistrian University of Athens
Locations (1):
- Department of Intensive Care Medicine Evaggelismos General Hospital, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ehler J, Barrett LK, Taylor V, Groves M, Scaravilli F, Wittstock M, Kolbaske S, Grossmann A, Henschel J, Gloger M, Sharshar T, Chretien F, Gray F, Noldge-Schomburg G, Singer M, Sauer M, Petzold A. Translational evidence for two distinct patterns of neuroaxonal injury in sepsis: a longitudinal, prospective translational study. Crit Care. 2017 Oct 23;21(1):262. doi: 10.1186/s13054-017-1850-7. PMID 29058589
- [Background] Taccone FS, Castanares-Zapatero D, Peres-Bota D, Vincent JL, Berre' J, Melot C. Cerebral autoregulation is influenced by carbon dioxide levels in patients with septic shock. Neurocrit Care. 2010 Feb;12(1):35-42. doi: 10.1007/s12028-009-9289-6. PMID 19806473
- [Background] Schramm P, Klein KU, Falkenberg L, Berres M, Closhen D, Werhahn KJ, David M, Werner C, Engelhard K. Impaired cerebrovascular autoregulation in patients with severe sepsis and sepsis-associated delirium. Crit Care. 2012 Oct 4;16(5):R181. doi: 10.1186/cc11665. PMID 23036135
- [Background] Bindra J, Pham P, Chuan A, Jaeger M, Aneman A. Is impaired cerebrovascular autoregulation associated with outcome in patients admitted to the ICU with early septic shock? Crit Care Resusc. 2016 Jun;18(2):95-101. PMID 27242107
- [Background] Donnelly J, Budohoski KP, Smielewski P, Czosnyka M. Regulation of the cerebral circulation: bedside assessment and clinical implications. Crit Care. 2016 May 5;20(1):129. doi: 10.1186/s13054-016-1293-6. PMID 27145751
- [Background] Wang D, Hu B, Hu C, Zhu F, Liu X, Zhang J, Wang B, Xiang H, Cheng Z, Xiong Y, Zhao Y, Li Y, Wang X, Peng Z. Clinical Characteristics of 138 Hospitalized Patients With 2019 Novel Coronavirus-Infected Pneumonia in Wuhan, China. JAMA. 2020 Mar 17;323(11):1061-1069. doi: 10.1001/jama.2020.1585. PMID 32031570
- [Background] Kaneko N, Satta S, Komuro Y, Muthukrishnan SD, Kakarla V, Guo L, An J, Elahi F, Kornblum HI, Liebeskind DS, Hsiai T, Hinman JD. Flow-Mediated Susceptibility and Molecular Response of Cerebral Endothelia to SARS-CoV-2 Infection. Stroke. 2021 Jan;52(1):260-270. doi: 10.1161/STROKEAHA.120.032764. Epub 2020 Nov 9. PMID 33161843
- [Background] Cagnazzo F, Piotin M, Escalard S, Maier B, Ribo M, Requena M, Pop R, Hasiu A, Gasparotti R, Mardighian D, Piano M, Cervo A, Eker OF, Durous V, Sourour NA, Elhorany M, Zini A, Simonetti L, Marcheselli S, Paolo NN, Houdart E, Guedon A, Ligot N, Mine B, Consoli A, Lapergue B, Cordona Portela P, Urra X, Rodriguez A, Bolognini F, Lebedinsky PA, Pasco-Papon A, Godard S, Marnat G, Sibon I, Limbucci N, Nencini P, Nappini S, Saia V, Caldiera V, Romano D, Frauenfelder G, Gallesio I, Gola G, Menozzi R, Genovese A, Terrana A, Giorgianni A, Cappellari M, Augelli R, Invernizzi P, Pavia M, Lafe E, Cavallini A, Giossi A, Besana M, Valvassori L, Macera A, Castellan L, Salsano G, Di Caterino F, Biondi A, Arquizan C, Lebreuche J, Galvano G, Cannella A, Cosottini M, Lazzarotti G, Guizzardi G, Stecco A, Tassi R, Bracco S, Bianchini E, Micieli C, Pascarella R, Napoli M, Causin F, Desal H, Cotton F, Costalat V; ET-COVID-19 Study Group*. European Multicenter Study of ET-COVID-19. Stroke. 2021 Jan;52(1):31-39. doi: 10.1161/STROKEAHA.120.031514. Epub 2020 Nov 23. PMID 33222617
- [Background] Alharthy A, Faqihi F, Papanikolaou J, Balhamar A, Blaivas M, Memish ZA, Karakitsos D. Thrombolysis in severe COVID-19 pneumonia with massive pulmonary embolism. Am J Emerg Med. 2021 Mar;41:261.e1-261.e3. doi: 10.1016/j.ajem.2020.07.068. Epub 2020 Jul 30. PMID 32763101
- [Background] Zangrillo A, Landoni G, Beretta L, Morselli F, Serpa Neto A, Bellomo R; COVID-BioB Study Group. Angiotensin II infusion in COVID-19-associated vasodilatory shock: a case series. Crit Care. 2020 May 15;24(1):227. doi: 10.1186/s13054-020-02928-0. No abstract available. PMID 32414393
- [Background] Dupont A, Rauch A, Staessens S, Moussa M, Rosa M, Corseaux D, Jeanpierre E, Goutay J, Caplan M, Varlet P, Lefevre G, Lassalle F, Bauters A, Faure K, Lambert M, Duhamel A, Labreuche J, Garrigue D, De Meyer SF, Staels B, Vincent F, Rousse N, Kipnis E, Lenting P, Poissy J, Susen S; Lille Covid Research Network (LICORNE). Vascular Endothelial Damage in the Pathogenesis of Organ Injury in Severe COVID-19. Arterioscler Thromb Vasc Biol. 2021 May 5;41(5):1760-1773. doi: 10.1161/ATVBAHA.120.315595. Epub 2021 Feb 25. PMID 33626910
- [Background] Ince C. The microcirculation is the motor of sepsis. Crit Care. 2005;9 Suppl 4(Suppl 4):S13-9. doi: 10.1186/cc3753. Epub 2005 Aug 25. PMID 16168069
- [Background] Donati A, Domizi R, Damiani E, Adrario E, Pelaia P, Ince C. From macrohemodynamic to the microcirculation. Crit Care Res Pract. 2013;2013:892710. doi: 10.1155/2013/892710. Epub 2013 Feb 27. PMID 23509621
- [Background] Salama C, Han J, Yau L, Reiss WG, Kramer B, Neidhart JD, Criner GJ, Kaplan-Lewis E, Baden R, Pandit L, Cameron ML, Garcia-Diaz J, Chavez V, Mekebeb-Reuter M, Lima de Menezes F, Shah R, Gonzalez-Lara MF, Assman B, Freedman J, Mohan SV. Tocilizumab in Patients Hospitalized with Covid-19 Pneumonia. N Engl J Med. 2021 Jan 7;384(1):20-30. doi: 10.1056/NEJMoa2030340. Epub 2020 Dec 17. PMID 33332779
- [Background] Jamil S, Mark N, Carlos G, Cruz CSD, Gross JE, Pasnick S. Diagnosis and Management of COVID-19 Disease. Am J Respir Crit Care Med. 2020 May 15;201(10):P19-P20. doi: 10.1164/rccm.2020C1. No abstract available. PMID 32223716
- [Background] Goodson CM, Rosenblatt K, Rivera-Lara L, Nyquist P, Hogue CW. Cerebral Blood Flow Autoregulation in Sepsis for the Intensivist: Why Its Monitoring May Be the Future of Individualized Care. J Intensive Care Med. 2018 Feb;33(2):63-73. doi: 10.1177/0885066616673973. Epub 2016 Oct 25. PMID 27798314
- [Background] Nakagawa I, Park HS, Yokoyama S, Yamada S, Motoyama Y, Park YS, Wada T, Kichikawa K, Nakase H. Indocyanine green kinetics with near-infrared spectroscopy predicts cerebral hyperperfusion syndrome after carotid artery stenting. PLoS One. 2017 Jul 12;12(7):e0180684. doi: 10.1371/journal.pone.0180684. eCollection 2017. PMID 28704454